CLINICAL TRIAL: NCT01188343
Title: Immunogenicity and Safety of Japanese Encephalitis Chimeric Virus Vaccine (JE CV) Concomitantly Administered With Measles, Mumps, and Rubella (MMR) Vaccine in Toddlers in Taiwan.
Brief Title: Study of Japanese Encephalitis Chimeric Virus Vaccine Given With Measles-Mumps-Rubella Vaccine in Taiwanese Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEC04; UTN: U1111-1112-2143 (Other: WHO)
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Japanese Encephalitis; Measles; Mumps; Rubella
Keywords: Japanese Encephalitis; Japanese encephalitis chimeric virus vaccine; Measles; Mumps; Rubella
MeSH Terms: conditions — Encephalitis, Japanese; Measles; Mumps; Rubella

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Participants will receive the Japanese encephalitis chimeric virus vaccine (JE-CV) on Day 0 and Measles, mumps, and rubella live attenuated virus vaccine (MMR) on Day 42
  Interventions: Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus
- Group 2 (Experimental): Participants will receive Measles, mumps, and rubella live attenuated virus vaccine (MMR) on Day 0, and the Japanese encephalitis chimeric virus vaccine (JE-CV) on Day 42.
  Interventions: Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus
- Group 3 (Experimental): Participants will receive the Measles, mumps, and rubella live attenuated virus vaccine (MMR) and the Japanese encephalitis chimeric virus vaccine (JE-CV) on Day 0
  Interventions: Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus

INTERVENTIONS:
Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus — 0.5 mL each; Subcutaneous (SC)
  Other Names: JE-CV; MMR II®
  Arms: Group 1
Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus — 0.5 mL each, Subcutaneous (SC)
  Other Names: JE-CV; MMR II®
  Arms: Group 2
Biological: Japanese encephalitis chimeric virus: Measles, mumps, and rubella live attenuated virus — 0.5 mL each, subcutaneous (SC)
  Other Names: JE-CV; MMR II®
  Arms: Group 3

SUMMARY:
This study is designed to compare the immunogenicity of Japanese encephalitis chimeric virus vaccine (JE-CV) and measles-mumps-rubella (MMR)vaccine when given together or when given at separate visits 6 weeks apart in toddlers aged 12 to 18 months.

Primary objective:

* To demonstrate the non-inferiority of the antibody responses in terms of seroconversion of the concomitant administration of JE-CV and MMR compared to the antibody responses after the single administration of JE-CV and MMR vaccine.

Secondary objectives:

* To describe the immune response to JE CV and MMR before and after one dose of JE CV and MMR vaccine, respectively.
* To describe the safety of a single dose of JE-CV and MMR vaccine (given separately at a 6-week interval and the safety of the concomitant administration of JE-CV and MMR vaccine in all subjects up to 6 months after last vaccination.

DETAILED DESCRIPTION:
All participants will receive Japanese encephalitis chimeric virus vaccine and measles-mumps-rubella vaccine and will be monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria

* Aged 12 to 18 months on the day of inclusion .
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg.
* Subject in good health based on medical history and physical examination.
* Provision of informed consent form signed by at least one parent or other legally acceptable representative, and by an independent witness if the parents or legally acceptable representative cannot read.
* Subject and parent/legally acceptable representative or delegate able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination except for pandemic influenza vaccination, which may be received at least two weeks before the study vaccines.
* Planned receipt of any vaccine up to the 6 weeks following the last trial vaccination except for pandemic influenza vaccine. In the event of a local or national immunization program with a pandemic influenza vaccine, participants who receive a pandemic influenza vaccine at any time during the trial will not be withdrawn from the trial.
* Previous vaccination against measles, measles-mumps-rubella (MMR), or flavivirus disease, including Japanese encephalitis (JE).
* Receipt of blood in the past 6 months that might interfere with the assessment of the immune response
* Receipt of intravenous injection of plasma, platelet product, or high dose of intravenous immunoglobulin in the past 11 months
* Receipt of intramuscular treatment of immunoglobulin or Hepatitis B immunoglobulin in the past 3 months
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known history of human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C seropositivity.
* History of measles, mumps, rubella, or flavivirus infection confirmed either clinically, serologically, or microbiologically.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing any of the same substances .
* Known systemic hypersensitivity to gelatin, eggs, or anaphylactic/anaphylactoid reaction to neomycin.
* Known history of thrombocytopenia.
* Administration of any anti-viral within 2 months preceding first vaccination and up to the 6 weeks following the last trial vaccination.
* History of central nervous system disorder or disease, including seizures and febrile seizures.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 542 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (3):
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan District

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 14 August 2010 through 28 July 2011 at 5 clinic centers in Taiwan.
Pre-assignment Details: A total of 550 participants who met all of the inclusion and none of the exclusion criteria were randomized, 542 were vaccinated and reported.
Groups:
- JE CV + MMR (Group 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE CV) on day 0 and one dose of Measles, Mumps, and Rubella (MMR) vaccine on day 42
- MMR + JE CV (Group 2): Participants 12 to 18 months of age received one dose of MMR vaccine on day 0 and one dose of JE CV vaccine on day 42
- JE CV/MMR (Group 3): Participants 12 to 18 months of age received one dose each of MMR and JE CV vaccine on day 0
Period: Overall Study
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Started | 102 | 219 | 221
Completed | 101 | 193 | 220
Not Completed | 1 | 26 | 1
Not completed — Not vaccinated | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 24 | 0

BASELINE CHARACTERISTICS:
Groups:
- JE CV/MMR (Group 3): Participants 12 to 18 months of age received one dose each of MMR and JE-CV vaccine on day 0
- Total: Total of all reporting groups
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3) | Total
Number analyzed (Participants) | 102 | 219 | 221 | 542
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 102 | 219 | 221 | 542
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.1 (1.12) | 13.0 (1.08) | 13.1 (1.19) | 13.1 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 110 | 109 | 265
  Male | 56 | 109 | 112 | 277
Region of Enrollment [Number; unit: Participants]
  Taiwan | 102 | 219 | 221 | 542

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion to Vaccine Antigens Following Concomitant Administration of Japanese Encephalitis Chimeric Virus Vaccine (JECV) and MMR or Single Administration of JE-CV and MMR Vaccine at 42 Days Following First Vaccination
Description: JE-CV antigens were measured using a 50% plaque reduction neutralization test (PRNT50); MMR antigens were measured using enzyme linked immunosorbent assay (ELISA). Seroconversion was defined as: for JE-CV - participants with a pre-vaccination titer <1/10 and post-vaccination titer ≥1/10, or a pre-vaccination titer ≥1/10 and 4-fold increase from pre- to post; for Measles - post-vaccination titer ≥120 mIU/ml, when pre-vaccination titer is <120 mIU/ml; for Mumps - post-vaccination titer ≥1/10 U/ml when pre-vaccination titer is <10 U/ml; and for Rubella, post-vaccination titer ≥1/10 U/ml when pre-vaccination titer is <10 U/ml.
Time Frame: Day 0 (pre-vaccination) and Day 42 post-vaccination
Population: Seroconversion was assessed in the Per Protocol Analysis Set with evaluable data.
Measure: Number; unit: Percentage of Participants
Groups:
- JE-CV + MMR (Group 1): Participants 12 to 18 months of age received one dose of Japanese encephalitis chimeric virus vaccine (JE-CV) on day 0 and one dose of Measles, Mumps, and Rubella (MMR) vaccine on day 42
- MMR + JE-CV (Group 2): Participants 12 to 18 months of age received one dose of MMR vaccine on day 0 and one dose of JE-CV vaccine on day 42
- JE-CV/MMR (Group 3): Participants 12 to 18 months of age received one dose each of MMR and JE-CV vaccine on day 0
Arm/Group | JE-CV + MMR (Group 1) | MMR + JE-CV (Group 2) | JE-CV/MMR (Group 3)
Number analyzed (Participants) | 95 | 176 | 197
Percentage of Participants
  JE-CV (N = 95, 0, 194) | 97.9 | NA [0 to 0] — JE-CV was not administered on Day 0 in this group | 96.9 [0 to 0]
  Measles (N = 0, 170, 193) | NA — MMR was not administered on Day 0 in this group. | 97.6 [0 to 0] | 100 [0 to 0]
  Mumps (N = 0, 173, 194) | NA — MMR was not administered on Day 0 in this group. | 98.8 [0 to 0] | 99.5 [0 to 0]
  Rubella (N = 0, 154, 178) | NA — MMR was not administered on Day 0 in this group. | 99.4 [0 to 0] | 99.4 [0 to 0]

2. Secondary Outcome: Percentage of Participants With Seroconversion to JE-CV and MMR Antigens Before and 42 Days Following Concomitant Administration of JE-CV and MMR or Single Administration of JE-CV and MMR Vaccine
Description: JE-CV antigens were measured using a 50% plaque reduction neutralization test (PRNT50); MMR antigens were measured using enzyme linked immunosorbent assay (ELISA). Seroconversion was defined as: for JE-CV - participants with a pre-vaccination titer <1/10 and post-vaccination titer ≥1/10, or a pre-vaccination titer ≥1/10 and 4-fold increase from pre- to post; for Measles - post-vaccination titer ≥120 mIU/ml, when pre-vaccination titer is <120 mIU/ml; for Mumps - post-vaccination titer ≥1/10 U/ml when pre-vaccination titer is <10 U/ml; and for Rubella, post-vaccination titer ≥1/10 U/ml when pre-vaccination titer is <10 U/m
Time Frame: Pre-vaccination and Day 42 post-vaccination
Population: Seroconversion to JE-CV and to MMR vaccine antigen was assessed in all participants who were randomized, vaccinated, who performed all protocol defined activities and has evaluable data (Per-protocol Analysis Set).
Measure: Number; unit: Percentage of Participants
Arm/Group | JE-CV + MMR (Group 1) | MMR + JE-CV (Group 2) | JE-CV/MMR (Group 3)
Number analyzed (Participants) | 95 | 176 | 197
Percentage of Participants
  JE-CV Pre-vaccination (N = 95, 158, 194) | 0.0 | 0.0 [0 to 0] | 0.0 [0 to 0]
  JE-CV Post-vaccination (N = 95, 158, 194) | 97.9 | 100.0 [0 to 0] | 96.9 [0 to 0]
  Measles Pre-vaccination (N = 94, 176, 196) | 4.3 | 2.8 [0 to 0] | 1.0 [0 to 0]
  Measles Post-vaccination (N = 94, 176, 197) | 97.9 | 97.7 [0 to 0] | 100.0 [0 to 0]
  Mumps Pre-vaccination (N = 94, 176, 196) | 1.1 | 1.1 [0 to 0] | 0.5 [0 to 0]
  Mumps Post-vaccination (N = 94, 176, 197) | 100.0 | 98.9 [0 to 0] | 99.5 [0 to 0]
  Rubella Pre-vaccination (N = 94, 176, 196) | 9.6 | 11.9 [0 to 0] | 8.7 [0 to 0]
  Rubella Post-vaccination (N = 94, 176, 197) | 100.0 | 99.4 [0 to 0] | 99.5 [0 to 0]

3. Secondary Outcome: Number of Participants With Seroprotection to JE-CV and MMR Antigens Before, at Month 6 After Last Vaccination and Month 12 After First Following Concomitant Administration of JE-CV and MMR or Single Administration of JE-CV and MMR Vaccine
Description: JE-CV antigens were measured using a 50% plaque reduction neutralization test (PRNT50); MMR antigens were measured using enzyme linked immunosorbent assay (ELISA). Seroprotection was defined as: for JE-CV - participants with a pre-vaccination titer <1/10 (1/dil) and post-vaccination titer ≥1/10, (1/dil) or a pre-vaccination titer ≥1/10 and 4-fold increase from pre- to post; for Measles - post-vaccination titer ≥120 mIU/ml, when pre-vaccination titer is <120 mIU/ml; for Mumps - post-vaccination titer ≥1/10 units/ml when pre-vaccination titer is <10 units/ml; and for Rubella, post-vaccination titer ≥1/10 IU/ml when pre-vaccination titer is <10 IU/m
Time Frame: Pre-vaccination and up to Month 12 post-vaccination
Population: Seroprotection to JE-CV and to MMR vaccine antigen was assessed in all participants who were randomized, vaccinated and who performed all protocol defined activities the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | JE-CV + MMR (Group 1) | MMR + JE-CV (Group 2) | JE-CV/MMR (Group 3)
Number analyzed (Participants) | 102 | 217 | 221
Participants
  JE-CV Pre-vaccination (N=102, 197, 221) | 2 | 10 | 4
  JE-CV 6 months Post-vaccination (N=96, 191, 217) | 92 | 190 | 203
  JE-CV 12 months Post-vaccination (N=89, 164, 193) | 86 | 162 | 171
  Measles Pre-vaccination (N = 101, 217, 219) | 4 | 8 | 2
  Measles 6 months Post-vaccination (N=96, 191, 217) | 93 | 189 | 216
  Measles 12 months Post-vaccination (N=89, 164, 193 | 87 | 163 | 192
  Mumps Pre-vaccination (N=101, 217, 219) | 1 | 2 | 2
  Mumps 6 months Post-vaccination (N=96, 191, 217) | 90 | 180 | 208
  Mumps 12 months Post-vaccination (N=89, 164, 193) | 82 | 153 | 176
  Rubella Pre-vaccination (N=101, 217, 219) | 10 | 23 | 19
  Rubella 6 months Post-vaccination (N=96, 191, 217) | 95 | 191 | 217
  Rubella 12 months Post-vaccination (N=89, 164, 193 | 89 | 164 | 192

4. Secondary Outcome: Geometric Mean Titers of Antibodies to Vaccine Antigens Before and After Concomitant Administration of JE-CV and MMR or Single Administration of JE-CV and MMR Vaccine
Description: JE-CV antigens were measured using a 50% plaque reduction neutralization test (PRNT50); MMR antigens were measured using enzyme linked immunosorbent assay (ELISA).
Time Frame: Pre-vaccination and Day 42 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set population with evaluable data.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Number analyzed (Participants) | 95 | 176 | 197
Titers
  JE-CV pre-vaccination (N = 95, 158, 194) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  JE-CV post-vaccination (N = 95, 158, 194) | 510 [356 to 731] | 581 [449 to 752] | 332 [258 to 426]
  Measles pre-vaccination (N = 94, 176, 196) | 34.3 [31.5 to 37.3] | 33.4 [31.4 to 35.5] | 33.4 [32.0 to 35.0]
  Measles post-vaccination (N = 94, 176, 197) | 1835 [1536 to 2193] | 1723 [1506 to 1971] | 1924 [1753 to 2111]
  Mumps pre-vaccination (N = 94, 176, 196) | 2.59 [2.46 to 2.71] | 2.63 [2.52 to 2.75] | 2.55 [2.49 to 2.62]
  Mumps Post-vaccination (N = 94, 176, 197) | 81.1 [70.1 to 93.9] | 87.5 [77.6 to 98.8] | 89.2 [80.0 to 99.5]
  Rubella pre-vaccination (N = 94, 176, 196) | 3.90 [3.44 to 4.43] | 3.97 [3.60 to 4.37] | 3.60 [3.32 to 3.90]
  Rubella post-vaccination (N = 94, 176, 197) | 78.0 [68.3 to 89.2] | 81.4 [73.7 to 89.9] | 69.6 [63.6 to 76.0]

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Administration of JE-CV Vaccine
Description: Solicited injection site: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Lost, and Irritability. Grade 3 injection site: Pain - Cries when injected limb is moved or movement of limb is reduced; Erythema and Swelling - ≥5 cm. Grade 3 systemic reactions: Fever - >39.5°C; Vomiting - ≥6 episodes per 24 hours or requiring parenteral hydration; Crying Abnormal - >3 hours; Drowsiness - Sleeping most of the time or difficult to wake; Appetite Lost - Refused ≥3 feeds/meals or refused most feeds/meals; Irritability - Inconsolable.
Time Frame: Day 0 up to Day14 post-vaccination
Population: Solicited injection site and systemic events were assessed in all randomized and vaccinated participants, the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Number analyzed (Participants) | 102 | 196 | 220
Participants
  Injection site Pain (N = 102, 195, 219) | 18 | 30 [0 to 0] | 35 [0 to 0]
  Grade 3 Pain (N = 102, 195, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema (N = 102, 195, 219) | 11 | 21 [0 to 0] | 24 [0 to 0]
  Grade 3 Erythema (N = 102, 195, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling (N = 102, 195, 219) | 2 | 11 [0 to 0] | 3 [0 to 0]
  Grade 3 Swelling (N = 102, 195, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Solicited Fever (N = 102, 195, 219) | 17 | 35 [0 to 0] | 53 [0 to 0]
  Grade 3 Fever (N = 102, 195, 219) | 1 | 1 [0 to 0] | 1 [0 to 0]
  Solicited Vomiting (N = 102, 195, 219) | 15 | 21 [0 to 0] | 39 [0 to 0]
  Grade 3 Vomiting (N = 102, 195, 219) | 0 | 3 [0 to 0] | 0 [0 to 0]
  Solicited Crying Abnormal (N = 102, 195, 219) | 24 | 56 [0 to 0] | 79 [0 to 0]
  Grade 3 Crying Abnormal (N = 102, 195, 219) | 2 | 4 [0 to 0] | 5 [0 to 0]
  Solicited Drowsiness (N = 102, 195, 219) | 26 | 45 [0 to 0] | 67 [0 to 0]
  Grade 3 Drowsiness (N = 102, 195, 219) | 0 | 3 [0 to 0] | 2 [0 to 0]
  Solicited Appetite Lost (N = 102, 195, 219) | 25 | 46 [0 to 0] | 78 [0 to 0]
  Grade 3 Appetite Lost (N = 102, 195, 219) | 3 | 5 [0 to 0] | 6 [0 to 0]
  Solicited Irritability (N = 102, 195, 219) | 28 | 39 [0 to 0] | 72 [0 to 0]
  Grade 3 Irritability (N = 102, 195, 219) | 4 | 0 [0 to 0] | 2 [0 to 0]

6. Other Pre Specified Outcome: Serological Status of Flavivirus at Before (Baseline) Concomitant Administration of JE-CV and MMR or Single Administration of JE-CV and MMR Vaccine
Description: Neutralizing antibodies levels against dengue were only evaluated on subjects ELISA positive for Immunoglobulin G (IgG) or Immunoglobulin M (IgM). Flavivirus positive was defined as antibodies against JE-CV virus ≥10 (l/dil) or antibodies against at least one dengue virus serotype ≥10 (l/dil); Flavivirus negative was defined as antibodies against JE CV virus < 10 (l/dil) and antibodies against the 4 dengue virus serotypes < 10 (l/dil).
Time Frame: Day 0 (pre-vaccination)
Population: Serological status of Flavivirus infection was assessed in the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Number analyzed (Participants) | 102 | 197 | 221
Participants
  JE-CV virus/dengue serotypes FV Positive | 2 | 18 [0 to 0] | 5 [0 to 0]
  JE CV virus/dengue serotypes FV Negative | 100 | 179 [0 to 0] | 216 [0 to 0]
  JE CV virus | 2 | 10 [0 to 0] | 4 [0 to 0]
  Any dengue serotype | 0 | 8 [0 to 0] | 1 [0 to 0]
  Dengue serotype 1 | 0 | 7 [0 to 0] | 1 [0 to 0]
  Dengue serotype 2 | 0 | 0 [0 to 0] | 0 [0 to 0]
  Dengue serotype 3 | 0 | 0 [0 to 0] | 0 [0 to 0]
  Dengue serotype 4 | 0 | 3 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Administration of MMR Vaccine
Description: as for outcome 5
Time Frame: Day 0 up to Day 14 post-vaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Number analyzed (Participants) | 101 | 219 | 220
Participants
  Injection site Pain (N = 101, 211, 219) | 16 | 32 [0 to 0] | 36 [0 to 0]
  Grade 3 Pain (N = 101, 211, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema (N = 101, 211, 219) | 7 | 22 [0 to 0] | 22 [0 to 0]
  Grade 3 Erythema (N = 101, 211, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling (N = 101, 211, 219) | 3 | 7 [0 to 0] | 4 [0 to 0]
  Grade 3 Swelling (N = 101, 211, 219) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Solicited Fever (N = 101, 211, 219) | 21 | 48 [0 to 0] | 53 [0 to 0]
  Grade 3 Fever (N = 101, 211, 219) | 1 | 4 [0 to 0] | 1 [0 to 0]
  Solicited Vomiting (N = 101, 210, 219) | 12 | 32 [0 to 0] | 39 [0 to 0]
  Grade 3 Vomiting (N = 101, 210, 219) | 0 | 2 [0 to 0] | 0 [0 to 0]
  Solicited Crying Abnormal (N = 101, 210, 219) | 30 | 73 [0 to 0] | 79 [0 to 0]
  Grade 3 Crying Abnormal (N = 101, 210, 219) | 4 | 7 [0 to 0] | 5 [0 to 0]
  Solicited Drowsiness (N = 101, 210, 219) | 26 | 68 [0 to 0] | 67 [0 to 0]
  Grade 3 Drowsiness (N = 101, 210, 219) | 1 | 4 [0 to 0] | 2 [0 to 0]
  Solicited Appetite Lost (N = 101, 210, 219) | 29 | 80 [0 to 0] | 78 [0 to 0]
  Grade 3 Appetite Lost (N = 101, 210, 219) | 0 | 10 [0 to 0] | 6 [0 to 0]
  Solicited Irritability (N = 101, 210, 219) | 26 | 64 [0 to 0] | 72 [0 to 0]
  Grade 3 Irritability (N = 101, 210, 219) | 4 | 3 [0 to 0] | 2 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Description: The total number (N) for solicited adverse events in the table reflects those participants for which the diary cards were returned and for which data were available for the event during the period.
Arm/Group | JE CV + MMR (Group 1) | MMR + JE CV (Group 2) | JE CV/MMR (Group 3)
Serious Adverse Events (participants affected / at risk) | 10/102 | 21/219 | 13/220
Other Adverse Events (participants affected / at risk) | 30/102 | 80/219 | 79/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE CV + MMR (Group 1) (N=102) | MMR + JE CV (Group 2) (N=219) | JE CV/MMR (Group 3) (N=220)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diarrhea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hand foot and mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 1 (1) | 5 (5) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | JE CV + MMR (Group 1) (N=102) | MMR + JE CV (Group 2) (N=219) | JE CV/MMR (Group 3) (N=220)
Somnolence (Nervous system disorders) | 26 (26) | 45/196 (45) | 67 (67)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2/196 (2) | 12 (12)
Injection site Pain (General disorders) | 18 (18) | 30/195 (30) | 35 (35)
Injection site Erythema (General disorders) | 11 (11) | 21/195 (21) | 24 (24)
Injection site Swelling (General disorders) | 2 (2) | 11/195 (11) | 3 (3)
Fever (General disorders) | 21/101 (21) | 48/211 (48) | 53 (53)
Vomiting (Gastrointestinal disorders) | 12/101 (12) | 32/210 (32) | 39 (39)
Crying Abnormal (Psychiatric disorders) | 30/101 (30) | 73/210 (73) | 79 (79)
Drowsiness (Nervous system disorders) | 26/101 (26) | 68/210 (68) | 67 (67)
Appetite Lost (Metabolism and nutrition disorders) | 29/101 (29) | 80/210 (80) | 78 (78)
Irritability (Psychiatric disorders) | 26/101 (26) | 64/210 (64) | 72 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.